CLINICAL TRIAL: NCT00055042
Title: Laser and Antioxidant Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030064; 03-EI-0064
Record Dates: First submitted 2003-02-15; First posted 2003-02-17 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-01

CONDITIONS: Macular Edema; Diabetes Mellitus
Keywords: Types 1 and 2 Diabetes; Diode Laser Photocoagulation; Vitamin E; Elevated Low-Density Lipoprotein (LDL-C) Cholesterol; Diabetes Type I; Diabetes Type II; Diabetic Macular Edema
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Vitamin E

INTERVENTIONS:
Drug: Vitamin E

SUMMARY:
This study will compare the side effects of two laser treatments for diabetic macular edema, a common condition in patients with diabetes. In macular edema, blood vessels in the retina-a thin layer of tissue that lines the back of the eye-become leaky and the retina swells. The macula-the center part of the retina that is responsible for fine vision-may also swell and cause vision loss. Traditional laser treatment (argon blue or green, or yellow) for macular swelling, or edema, causes scarring that can expand and possibly lead to more loss of vision. A different type of laser (diode) may have less damaging effects to the eye and fewer long-term adverse effects, but this is not known. The results of this study on side effects of the treatments will be used to design a larger study of effectiveness. The study will also examine whether vitamin E can reduce the damage caused by laser treatment. Patients with elevated cholesterol levels will be invited to participate in a cholesterol reduction part of the study to compare normal-pace cholesterol reduction with accelerated reduction.

Patients 18 years of age and older with type 1 or type 2 diabetes and macular edema may be eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history and physical examination.
* Eye examination to assess visual acuity (eye chart test) and eye pressure, and to examine pupils, lens, retina and eye movements. The pupils will be dilated with drops for this examination.
* Blood tests to measure cholesterol and vitamin E blood levels, blood clotting time, hemoglobin A1C (a measure of diabetes control), and to evaluate liver and kidney function.
* Eye photography to help evaluate the status of the retina and changes that may occur in the future. Special photographs of the inside of the eye are taken using a camera that flashes a bright light into the eye.
* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Multifocal electroretinogram to measure electrical responses generated within the retina. The test, which takes about 1-1/2 hours, is painless.

Participants will be randomly assigned to take 1600 IU of vitamin E or placebo (an inactive, look-alike pill) daily. After taking the pills for 3 months or more, patients who require laser treatment will be randomly assigned to one of the two laser therapies. (Patients with macular edema in both eyes will receive both treatments, one in each eye.) For these procedures, eye drops are put in the eye to numb the surface and a contact lens is placed on the eye during the laser beam application. Several visits may be required for additional laser treatments. The maximum number of treatments depends on how well they are working. Patients will return for follow-up visits 1, 3, and 6 months after the first treatment, and then every 6 months until either the patient returns for a 3-year visit; the last enrolled patient returns for the 1-year visit; or the patient requests to leave the study. During the follow-up visits, patients' response to treatment will be evaluated with repeat tests of several of the screening exams.

DETAILED DESCRIPTION:
This randomized pilot study is an important first step in planning a large multi-center clinical trial to evaluate medical and laser approaches that could improve the visual outcome for patients with diabetic retinopathy. This study will provide preliminary safety and efficacy data on these therapies as well as allow for assessment of the performance of ocular outcomes and study design for use in subsequent trials. If there are no safety concerns, the results of this pilot will be helpful in the design of a large multicenter clinical trial by providing data on estimates of expected treatment effects.

Using a factorial design, this study will compare (1) photocoagulation using a diode (micropulse) laser to mild Early Treatment Diabetic Retinopathy Studt (ETDRS) style (continuous wave laser using green or yellow wavelength) focal photocoagulation and, (2) the effect of treating with antioxidants (high dose Vitamin E) to placebo prior to and following laser photocoagulation. The primary outcome is a visual acuity drop or increase of 15 letters or more from baseline three year after enrollment. The secondary outcomes will be a 50% reduction in retinal thickening as measured by Optical Cohenrence Tomography (OT), a two-step reduction in macular thickness when compared to standard stereoscopic fundus photographs, and a 50% reduction in the area of leakage as measured by fluorescein angiography at 1 year amd 3 years after the initial laser compared to baseline. Additional outcomes will include the time (from baseline) of the first laser treatment and the number of retreatments required during the course of the study. These outcomes will be assessed for potential use in future trials. We are concerned with the following specific questions regarding safety and efficacy:

Safety

Is the risk of visual loss in patients with clinically significant diabetic macular edema potentially different across treatment groups?

Efficacy

Is there any evidence that any treatment combinations could be effective in reducing retinal thickening?

Is there any evidence that Vitamin E may affect the ability of either photocoagulation method to reduce retinal thickening, or vice versa?

What are the estimated treatment effects on vision?

Is the number of laser treatments required to achieve a reduction in retinal thickening similar across treatment groups?

A tertiary objective of this study will be to examine the effects of dramatically reducing low-density lipoproteins cholesterol in patients with diabetic macular edema and elevated serum lipids. Change in vision and change in retinal thickness will be compared across three groups; (1) patients who do not have elevated serum lipids at baseline, (2) patients who have elevated lipids at baseline and receive standard of care treatment, and (3) patients who have elevated lipids at baseline and are aggressively treated pharmacologically. This tertiary objective will be assessed for the feasibility of this randomization.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients with type 1 or 2 diabetes.
2. Patients with clinically significant macular edema in at least one eye.
3. Best corrected visual acuity 20/400 or better as measured on an ETDRS chart in the eye(s) with clinically significant macular edema.
4. May have had proliferative diabetic retinopathy but scatter photocoagulation must be performed more than six months ago.
5. Ocular media sufficiently clear to allow for quality fundus photography.
6. If aphakic or pseudophakic, lens removal must have occurred at least 6 months prior to enrollment.
7. Patient's medical status must include a likelihood of survival for 5 years.
8. Willingness to accept randomization for diet or drug therapy for lowering of elevated lipid levels.
9. Understand and sign the informed consent.
10. Patients over 18 years of age since the population of interest is primarily older than 18.

EXCLUSION CRITERIA:

1. Retinopathy that requires scatter photocoagulation immediately.
2. Ocular disease other than diabetic retinopathy that may confound the outcome of the study (e.g. age-related macular degeneration, drug toxicity, uveitis, etc.).
3. Poor likelihood of survival (of one year) due other systemic diseases (separate from diabetes).
4. Poor glycemic control with hemoglobin A1C greater than 12% within one month of baseline.
5. Past or current liver disease, which precludes the use of the lipid-lowering drugs.
6. Vitamine E supplementation over and above the amount in a myltivitamin (60 IU/day) one month prior to entry into the study.
7. History of hypersensitivity to fluorescein.
8. Prior or current macular detachment in the eligible eye(s).
9. Concurrent coumadin therapy or known bleeding diathesis.
10. Concurrent lithium therapy.
11. Concurrent treatment with a new investigational drug.
12. Malabsorption syndrome.
13. Concurrent administration of the anti-obesity drug orlistat Xenical).
14. Pregnant or lactating women.
15. Chronic requirement for any ocular medication for diseases that in the judgement of the examining physician, are vision threatening or may affect the primary outcome.
16. Current history of malignancy (except participants having a basal cell carcinoma that was treated successfully, or other malignancy operated on and in remission for 5 years prior to inclusion in the trial).
17. Participants whose diabetic macular edema, in the opinion of the Principal Investigator, cannot benefit from laser treatments, including those with subretinal fibrosis, severe macular non-perfusion, or parafoveal leakage in both eyes.
18. Participants that have a history of focal laser treatment, and are thought to be refractory to laser treatment or were treated within 3 months of baseline. (a minimal number of previous laser treatments are acceptable at the discretion of the Investigator.)
19. Participants with clear vitreal-retinal traction in both eyes.
20. Participants requiring therapy with topical prostaglandin analogues.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-02; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Klein BE, Moss SE, Klein R, Surawicz TS. The Wisconsin Epidemiologic Study of Diabetic Retinopathy. XIII. Relationship of serum cholesterol to retinopathy and hard exudate. Ophthalmology. 1991 Aug;98(8):1261-5. doi: 10.1016/s0161-6420(91)32145-6. PMID 1923364
- [Background] Lewis H, Schachat AP, Haimann MH, Haller JA, Quinlan P, von Fricken MA, Fine SL, Murphy RP. Choroidal neovascularization after laser photocoagulation for diabetic macular edema. Ophthalmology. 1990 Apr;97(4):503-10; discussion 510-1. doi: 10.1016/s0161-6420(90)32574-5. PMID 1691477
- [Background] Han DP, Mieler WF, Burton TC. Submacular fibrosis after photocoagulation for diabetic macular edema. Am J Ophthalmol. 1992 May 15;113(5):513-21. doi: 10.1016/s0002-9394(14)74722-1. PMID 1575225